CLINICAL TRIAL: NCT07039240
Title: Short-Term Effects of Trigger Point Dry Needling on Neuromuscular Control in Individuals Following Anterior Cruciate Ligament Reconstruction: A Single-Blind Randomized Controlled Trial
Brief Title: Short-Term Effects of Trigger Point Dry Needling on Neuromuscular Control in Individuals Following Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Ricardo Paredes, PhD Student, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1804202211322
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Knee; Anterior cruciate ligament; Neuromuscular control; Electromyography
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Dry Needling (Experimental)
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — The dry needling intervention will follow the fast-in and fast-out technique using disposable stainless-steel needles (0.35 × 40 mm). After insertion with a quick thrust, the needle will be manipulated in multiple directions to elicit at least one local twitch response (LTR). Once the first LTR is obtained, the needle will be moved vertically within a range of 3-5 mm, without rotation, until a total of three LTRs are elicited. The intervention is expected to last approximately 25-30 seconds.
  Arms: Dry Needling

SUMMARY:
This single-blind, randomized controlled trial aims to investigate the effects of dry needling on neuromuscular control in individuals with anterior cruciate ligament reconstruction during a single-leg vertical drop landing task. Participants in the intervention group will receive dry needling, while those in the control group will not receive any therapeutic intervention.

The main research question is:

• Can dry needling induce changes in muscle activation, co-contraction magnitude, and biomechanical parameters during landing?

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have undergone anterior cruciate ligament reconstruction
* Successful return to recreational sports participation
* For the experimental group, participants must present at least one active or latent trigger point in the vastus medialis (VM) and/or vastus lateralis (VL) muscles on the side ipsilateral to the ligament reconstruction.

Exclusion Criteria:

* Peripheral or central neurological disorders
* Systemic or degenerative diseases
* Fibromyalgia
* Iron deficiency
* Hypothyroidism
* Belonephobia
* Contraindications to dry needling
* History of dry needling treatment in the lower limbs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Co-contraction Index | Outcome measures will be assessed at baseline and 10 minutes post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Rehabilitation Research (CIR), School of Health of Polytechnic of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided